CLINICAL TRIAL: NCT02413489
Title: An Open Label, Phase 2 Study to Evaluate Efficacy and Safety of Daratumumab in Relapsed or Refractory Mantle Cell Lymphoma, Diffuse Large B-Cell Lymphoma, and Follicular Lymphoma
Brief Title: An Efficacy and Safety Proof of Concept Study of Daratumumab in Relapsed/Refractory Mantle Cell Lymphoma, Diffuse Large B-Cell Lymphoma, and Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DLBCL and FL cohorts met the pre-specified futility criteria and will not proceed. The MCL cohort was terminated due to slow recruitment and aggressive disease.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR106660; 54767414LYM2001 (Other: Janssen Research & Development, LLC); 2014-005299-26 (EudraCT Number)
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular
Keywords: Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Daratumumab
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): Participants will receive daratumumab (16 milligram per kilogram [mg/kg]) as intravenous infusion once every week for 8 weeks; then once every other week for 16 weeks; thereafter once every 4 weeks until documented progression, unacceptable toxicity, or study end.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab 16 mg/kg will be administered as intravenous infusion to participants once every week for 8 weeks; then once every other week for 16 weeks; thereafter once every 4 weeks until documented progression, unacceptable toxicity, or study end.

SUMMARY:
The purpose of this study is to assess overall response rate [ORR, including complete response (CR) and partial response (PR)], of daratumumab in participants with non-Hodgkin's lymphoma [a cancer of the lymph nodes (or tissues)-NHL] and to evaluate association between ORR and CD38 expression level in order to determine a threshold for CD38 expression level in each NHL subtype, above which daratumumab activity is enhanced in participants with relapsed or refractory mantle cell lymphoma, diffuse large B-cell lymphoma, and follicular lymphoma.

DETAILED DESCRIPTION:
This is an open label (everyone knows the study intervention), Phase 2 study to evaluate efficacy and safety of daratumumab in relapsed or refractory mantle cell lymphoma, diffuse large B-cell lymphoma, and follicular lymphoma. The study will have three phases. Screening phase, treatment phase, follow-up phase. Participants will receive daratumumab (16 milligram per kilogram [mg/kg]) as intravenous infusion approximately 3.5 years. Participants will primarily be assessed for overall response rate. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Has diagnosis and prior treatment for each non-hodgkin's lymphoma (NHL) subtype as defined below: Mantle cell lymphoma (MCL): pathologically verified diagnosis of MCL based on local pathology report, relapsed or refractory disease after at least 2 prior lines of therapy, including at least 1 cycle of Bruton's tyrosine kinase (BTK) inhibitor therapy and documented progressive disease (PD) during or after BTK inhibitor treatment or participants who could not tolerate BTK inhibitor [ie, discontinued BTK inhibitor due to adverse events (AEs)], b) Diffuse large B cell lymphoma (DLBCL): pathologically confirmed diagnosis of non-transformed DLBCL, and relapsed or refractory disease; for those participants who have not received HDT/ASCT are not eligible for HDT/ASCT due to comorbidities, c) Follicular lymphoma (FL): pathologically confirmed diagnosis of FL of Grade 1, 2, or 3a according to World Health Organization (WHO) criteria without pathological evidence of transformation, and relapsed disease after at least two prior systemic therapies including one anti-CD20 containing combination regimen
* At least 1 measurable site of disease
* Participants must have available archival or fresh tumor tissue or both to submit to a central laboratory for CD38 assay. Expression of CD38 is measured by immunohistochemistry on fresh or archived tumor sample by central assessment using a CD38 investigational IHC assay under development: a) Stage 1: participants whose tumors are more than or equal to (>=) 50 percent (%) positive for CD38, b) Stage 2: participant has less than (<) 50% CD38+ or greater than (>) 50% CD38+ depending on the distribution of CD 38 expression of enrolled participants during Stage 2. The sponsor will advise on which eligibility criterion is permitted during the enrollment period
* Participant must have an ECOG performance status score of 0 or 1
* Women of childbearing potential must be practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for participants participating in clinical studies: example, established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization (the vasectomized partner should be the sole partner for that participant); true abstinence (when this is in line with the preferred and usual lifestyle of the participant) during and after the study (3 months after the last dose of any component of the treatment regimen)
* A woman of childbearing potential must have a negative serum or urine pregnancy test within 14 days before commencing treatment. Females of reproductive potential must commit either to abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control example, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of any component of the treatment regimen. The exception to this restriction is that if the participant's female partner is surgically sterile, a second method of birth control is not required

Exclusion Criteria:

* Known central nervous system lymphoma
* Prior anti-tumor therapy including (all times measured prior to start of study drug): nitrosoureas within 6 weeks, chemotherapy within 3 weeks, therapeutic antibodies within 4 weeks, radio- or toxin-immunoconjugates within 10 weeks, radiation therapy within 2 weeks, investigational agents within 3 weeks, unless antibody this should be within 4 weeks
* Daratumumab or other anti-CD38 therapies
* Participant has a history of malignancy (other than NHL) within 3 years before the screening period (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, non-muscle invasive bladder cancer (papillary neoplasms of low malignant potential and primary non-invasive tumors), or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 2 years)
* Participant has known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) less than (<) 50% predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 <50% b) Participant has known moderate or severe persistent asthma within 2 years (see Attachment 4: NHLBI table of asthma severity), or currently has uncontrolled asthma of any classification. (Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (35):
- United States (14):
  - Duarte, California
  - Fountain Valley, California
  - Jacksonville, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Rochester, Minnesota
  - Omaha, Nebraska
  - New Brunswick, New Jersey
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Seattle, Washington
- Australia (3):
  - Adelaide
  - Box Hill
  - Melbourne
- Belgium (2):
  - Bruges
  - Ghent
- France (7):
  - Lille
  - Limoges
  - Nantes
  - Paris
  - Pessac
  - Pierre-Bénite
  - Rouen
- Netherlands (3):
  - Amsterdam
  - Rotterdam
  - Utrecht
- South Korea (2):
  - Goyang-si
  - Seoul
- Turkey (Türkiye) (4):
  - Ankara
  - Atakum
  - Istanbul
  - Kocaeli

REFERENCES:
- [Derived] Salles G, Gopal AK, Minnema MC, Wakamiya K, Feng H, Schecter JM, Wang M. Phase 2 Study of Daratumumab in Relapsed/Refractory Mantle-Cell Lymphoma, Diffuse Large B-Cell Lymphoma, and Follicular Lymphoma. Clin Lymphoma Myeloma Leuk. 2019 May;19(5):275-284. doi: 10.1016/j.clml.2018.12.013. Epub 2019 Jan 2. PMID 30795996

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total 36 participants were treated (15 participants in the diffuse large B-cell lymphoma [DLBCL] cohort, 16 participants in the follicular lymphoma [FL] cohort, and 5 participants in the mantle cell lymphoma [MCL] cohort).
Groups:
- Diffuse Large B-cell Lymphoma (DLBCL): Participants received daratumumab 16 milligram per kilogram (mg/kg) as intravenous infusion once every week for 8 weeks, then once every other week for 16 weeks, thereafter once every 4 weeks until documented progression, unacceptable toxicity or study end.
- Follicular Lymphoma (FL); Mantle Cell Lymphoma (MCL): Participants received daratumumab 16 mg/kg as intravenous infusion once every week for 8 weeks, then once every other week for 16 weeks, thereafter once every 4 weeks until documented progression, unacceptable toxicity or study end.
Period: Overall Study
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Mantle Cell Lymphoma (MCL)
Started | 15 | 16 | 5
Completed | 0 | 0 | 0
Not Completed | 15 | 16 | 5
Not completed — Death | 11 | 3 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Study Terminated By Sponsor | 2 | 13 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Mantle Cell Lymphoma (MCL) | Total
Number analyzed (Participants) | 15 | 16 | 5 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 4 | 18
  >=65 years | 10 | 7 | 1 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (11.88) | 62.3 (9.77) | 59.8 (6.69) | 63.8 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 0 | 11
  Male | 9 | 11 | 5 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 12 | 15 | 2 | 29
  Unknown or Not Reported | 3 | 0 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 2 | 0 | 6
  White | 7 | 13 | 2 | 22
  Unknown | 1 | 0 | 0 | 1
  Not Reported | 3 | 1 | 1 | 5
  Other | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 0 | 2 | 0 | 2
  Belgium | 2 | 0 | 0 | 2
  France | 4 | 2 | 0 | 6
  Netherlands | 2 | 3 | 2 | 7
  Republic of Korea | 4 | 2 | 0 | 6
  Turkey | 2 | 2 | 1 | 5
  United States | 1 | 5 | 2 | 8
CD38 expression value [Mean (Standard Deviation); unit: Percentage of CD38 expression] — The expression levels of CD38 were used to do diagnosis of MCL, DLBCL, or FL and measurable disease.
  Percentage of CD38 expression | 76.3 (18.07) | 70.3 (16.78) | 64 (8.22) | 71.9 (16.66)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved complete response (CR) or partial response (PR). As per Revised Response Criteria for Malignant Lymphoma, Lymph node measurements were taken from Computed Tomography (CT), CT portion of the Positron Emission Tomography/Computed Tomography (PET/CT), or Magnetic resonance imaging (MRI) scans where applicable. CR is defined as complete disappearance of all evidence of disease; PR as a greater than (>) 50 percent (%) decrease in the sum of the products of the maximal perpendicular diameters of measured lesions (SPD) and no new sites.
Time Frame: After the first dose until disease progression, withdrawal of consent from study participation, or the end of study (approximately 1.9 years)
Population: The analysis population was all participants that were treated with daratumumab.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Mantle Cell Lymphoma (MCL)
Number analyzed (Participants) | 15 | 16 | 5
Percentage of participants | 6.7 [0.2 to 31.9] | 12.5 [1.6 to 38.3] | 0 [NA to NA] — Confidence interval was not estimable as no participants had response.

2. Secondary Outcome: Duration of Response
Description: Duration of response was the duration from the date of the initial documentation of a response to the date of first documented evidence of progressive disease (PD). PD is defined as any new lesion >1.5 centimeter (cm) in any axis or greater than or equal to (>=) 50% increase in previously involved sites.
Time Frame: Approximately 1.9 years
Population: The analysis population was all participants that were treated with daratumumab and who achieved overall response There was insufficient data to perform Kaplan Meier analysis, therefore individual data for each evaluable participant was reported.
Measure: Number; unit: Months
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Mantle Cell Lymphoma (MCL)
Number analyzed (Participants) | 1 | 2 | 0
Months
  Participant 1 | 1.6 | 0.7 |
  Participant 2 | NA — Only 1 participant achieved response in DLBCL group. | 7.4 |

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the duration from the date of the first daratumumab dose to the date of progression or death, whichever comes first.
Time Frame: Approximately 1.9 years
Population: The analysis population was all participants that were treated with daratumumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Mantle Cell Lymphoma (MCL)
Number analyzed (Participants) | 15 | 16 | 5
Months | 1.2 [0.6 to 1.7] | 3.3 [1.9 to 3.8] | 1.3 [0.5 to 1.9]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the duration from the date of the first daratumumab dose to the date of death.
Time Frame: Approximately 1.9 years
Population: The analysis population was all participants that were treated with daratumumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Mantle Cell Lymphoma (MCL)
Number analyzed (Participants) | 15 | 16 | 5
Months | 4.9 [2.1 to 9.0] | 17.2 [15.0 to NA] — NA indicates upper limit of Confidence Interval was not estimable due to less number of participants with events. | 4.8 [1.7 to NA] — Upper limit of CI could not be estimated due to less number of participants analyzed.

5. Secondary Outcome: Time to Response
Description: Time to response was defined as the duration from the date of the first dose of daratumumab to the earliest date that a response (CR/PR) is first documented.
Time Frame: Approximately 1.9 years
Population: as for outcome 2
Measure: Number; unit: Months
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Mantle Cell Lymphoma (MCL)
Number analyzed (Participants) | 1 | 2 | 0
Months
  Participant 1 | 1.9 | 2.3 |
  Participant 2 | NA — Only 1 participant achieved response in DLBCL group. | 1.9 |

ADVERSE EVENTS:
Time Frame: Up to 1.9 years
Description: Analysis set included all participants who received at least 1 dose of study treatment and contributed any safety data after the start of study treatment.
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Mantle Cell Lymphoma (MCL)
All-Cause Mortality (participants affected / at risk) | 11/15 | 3/16 | 4/5
Serious Adverse Events (participants affected / at risk) | 6/15 | 6/16 | 3/5
Other Adverse Events (participants affected / at risk) | 15/15 | 16/16 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-cell Lymphoma (DLBCL) (N=15) | Follicular Lymphoma (FL) (N=16) | Mantle Cell Lymphoma (MCL) (N=5)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 0
Pneumonia Cytomegaloviral (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-cell Lymphoma (DLBCL) (N=15) | Follicular Lymphoma (FL) (N=16) | Mantle Cell Lymphoma (MCL) (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymph Node Pain (Blood and lymphatic system disorders) | 2 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 2 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Erythema of Eyelid (Eye disorders) | 0 | 1 | 0
Eyelid Oedema (Eye disorders) | 0 | 1 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 1 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 5 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1 | 0
Anal Incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 2
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 1 | 0
Swollen Tongue (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Catheter Site Erythema (General disorders) | 1 | 0 | 0
Catheter Site Inflammation (General disorders) | 1 | 0 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0
Chills (General disorders) | 2 | 1 | 1
Fatigue (General disorders) | 4 | 3 | 1
General Physical Health Deterioration (General disorders) | 1 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 2 | 0
Malaise (General disorders) | 3 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 1
Oedema Peripheral (General disorders) | 1 | 2 | 1
Pain (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 2 | 4 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Genital Herpes (Infections and infestations) | 0 | 1 | 0
Groin Infection (Infections and infestations) | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 3 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 2 | 0 | 0
C-Reactive Protein Increased (Investigations) | 1 | 0 | 0
Cytomegalovirus Test Positive (Investigations) | 1 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 1 | 1 | 0
Prostatic Specific Antigen Increased (Investigations) | 0 | 1 | 0
Weight Decreased (Investigations) | 3 | 2 | 0
Weight Increased (Investigations) | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Peripheral Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 5 | 1
Nerve Compression (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 0 | 1 | 0
Sensory Disturbance (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Thrombosis in Device (Product Issues) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depressed Mood (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urine Flow Decreased (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Oropharyngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blood Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Flushing (Vascular disorders) | 0 | 2 | 1
Hot Flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 3 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to 2 non-Hodgkin's lymphoma (NHL) sub types (DLBCL and FL cohorts) meeting the futility criteria defined in the protocol and the MCL cohort not having adequate recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-01-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT02413489/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT02413489/SAP_001.pdf